CLINICAL TRIAL: NCT04708054
Title: Venetoclax to Improve Outcomes of Fractionated Busulfan Regimen in Patients With High-Risk AML and MDS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0790; NCI-2020-13919 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0790 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Busulfan; Cladribine; fludarabine phosphate; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Thiotepa; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, busulfan, fludarabine, cladribine) (Experimental): Patients receive venetoclax PO QD on days -22 to -3, busulfan IV over 3 hours on days -20, -13, -6, -5, -4, and -3, and fludarabine phosphate IV over 1 hour and cladribine IV over 2 hours on days -6 to -3 in the absence of disease progression or unacceptable toxicity. Patients then undergo stem cell transplantation over 1-2 hours on day 0.
  Interventions: Drug: Busulfan; Drug: Cladribine; Drug: Fludarabine Phosphate; Procedure: Hematopoietic Cell Transplantation; Drug: Thiotepa; Drug: Venetoclax

INTERVENTIONS:
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Procedure: Hematopoietic Cell Transplantation — Undergo stem cell transplantation
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; Stem Cell Transplant; stem cell transplantation
Drug: Thiotepa — Given IV
  Other Names: 1,1'',1''''-Phosphinothioylidynetrisaziridine; Girostan; N,N'', N''''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies the effect of venetoclax together with busulfan, cladribine, and fludarabine in treating patients with high-risk acute myeloid leukemia or myelodysplastic syndrome who are undergoing stem cell transplant. Chemotherapy drugs, such as venetoclax, busulfan, cladribine, and fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Adding venetoclax to the current standard of care stem cell transplant regimen of busulfan, fludarabine, and cladribine may help to control high-risk acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
Phase 2 Portion

Primary Objective 1) To obtain preliminary evidence of efficacy as defined by 1-year progression free survival.

Secondary Objectives

To determine:

1. Safety of this regimen as per NCI toxicity criteria
2. Time to neutrophil and platelet engraftment
3. Incidence of acute and chronic GVHD
4. Relapse incidence
5. Non-relapse mortality
6. Overall survival
7. Graft versus host disease-relapse free survival (GRFS)

Phase 3 Portion

Primary Objective

1) To compare progression free survival between two arms Arm 1 Standard of Care: fludarabine + IV busulfan (FluBu) versus Arm 2 Experimental: Venetoclax + Fractionated busulfan, cladribine, and fludarabine

Secondary Objectives To compare following between two arms

1. Safety of this regimen as per NCI toxicity criteria
2. Time to neutrophil and platelet engraftment
3. Incidence of acute and chronic GVHD
4. Relapse incidence
5. Non-relapse mortality
6. Overall survival
7. Graft versus host disease-relapse free survival (GRFS)

ELIGIBILITY:
Inclusion Criteria:

Phase II

1. Age ≥ 18 and ≤ 70 years. English and non-English speaking patients are eligible.
2. Patients with acute myeloid leukemia who have previously received induction therapy and one of the following high-risk features:

   1. ELN17 adverse risk prognostic group irrespective of remission status (see Appendix 2)
   2. Measurable residual disease positive (MRD +)
   3. Not in complete remission including complete remission without count recovery (Cri) and/or morphologic leukemia free state (MLFS), primary refractory, or relapsed disease. See Appendix 3 for details.
   4. AML secondary to MDS or MPD
   5. Therapy-related AML.
   6. Not in complete remission after one course of induction therapy

   Or

   Patients with myelodysplastic syndrome or CMML and one of the following high-risk features:
   1. Poor or Very poor cytogenetic risk group as per IPSS-R
   2. Mutated P53 or Ras pathway genes (CBL, NRAS, KRAS, NF1, PTPN1) or DNMT 3a or ASXL1 or RUNX1
   3. Maximum IPSS-R >3.5 between diagnosis and the start of the preparative regimen.
   4. ≥ 5% BM blasts at transplant
   5. Therapy-related MDS
3. HLA-identical sibling or a minimum of 7/8 matched unrelated donor, or a haploidentical related donor available
4. Subject must voluntarily sign an informed consent
5. Female subjects of childbearing potential must have negative results for pregnancy test
6. Adequate hepatic and renal function per local laboratory reference range as follows:

   * Aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0X ULN
   * Bilirubin <1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
   * Subject must have adequate renal function as demonstrated by a creatinine clearance ≥ 50 mL/min; calculated by the Cockcroft Gault formula or measured by 24 hours urine collection.

Phase III

1. Age ≥ 18 and ≤ 65 years. English and non-English speaking patients are eligible.
2. Patients with acute myeloid leukemia who have previously received induction therapy and one of the following high-risk features:

   1. ELN22 adverse risk prognostic group irrespective of remission status (see Appendix
   2. Measurable residual disease positive (MRD +) including MRD + any time after induction therapy.
   3. Not in complete remission including complete remission without count recovery (Cri) and/or morphologic leukemia free state (MLFS), primary refractory, or relapsed disease. See Appendix 4 for details.
   4. AML secondary to MDS or MPD
   5. Therapy-related AML.
   6. Not in complete remission after one course of induction therapy
   7. Second or higher complete remission

   Or

   Patients with myelodysplastic syndrome and one of the following high-risk features:
   1. Poor or Very poor cytogenetic risk group as per IPSS-R
   2. Mutated P53 or Ras pathway genes (CBL, NRAS, KRAS, NF1, PTPN11) or ASXL1 or RUNX1 or moderate high, or high, or very high-risk group as per IPSS-M
   3. Maximum IPSS-R >3.5 between diagnosis and the start of the preparative regimen.
   4. ≥ 5% BM blasts at transplant
   5. Therapy-related MDS

   Or

   Patients with CMML
3. HLA-identical sibling or a minimum of 7/8 matched unrelated donor
4. Subject must voluntarily sign an informed consent
5. Female subjects of childbearing potential must have negative results for pregnancy test
6. Adequate hepatic and renal function per local laboratory reference range as follows:

   * Aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0X ULN
   * Bilirubin <1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
   * Subject must have adequate renal function as demonstrated by a creatinine clearance ≥ 50 mL/min; calculated by the Cockcroft Gault formula or measured by 24 hours urine collection.

Exclusion criteria:

1. Subject is known to be positive for HIV.
2. Subject has cognitive impairments and/or is a prisoner.
3. Subject has acute promyelocytic leukemia
4. Subject has known active CNS involvement with AML.
5. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

   1. Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
   2. Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.
6. Cardiac history of CHF requiring treatment or Ejection Fraction < 50% or unstable angina;
7. Corrected DLCO < 50% or FEV1 <65%.
8. Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

   * grapefruit or grapefruit products
   * Seville oranges (including marmalade containing Seville oranges)
   * star fruit
9. Patients with cognitive impairments and/or any serious unstable pre-existing medical condition or psychiatric disorder that can interfere with safety or with obtaining informed consent or compliance with study procedures.
10. Prior allogeneic stem cell transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year progression free survival (PFS) | At 1 year post-transplant
  The proportion of patients who are alive without disease relapse (PFS) at one year will be reported along with the corresponding 95% credible interval. Cox proportional hazards regression will be used to assess the association between PFS and clinical and treatment covariates of interest.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 3 years post-transplant
  OS will be calculated from the time of transplant by the method of Kaplan and Meier.
Graft-versus (vs.)-host disease-free, relapse-free survival (GRFS) | Up to 3 years post-transplant
  GRFS will be calculated from the time of transplant by the method of Kaplan and Meier.
Time to platelet engraftment | From the time of transplant up to 3 years
  The time to platelet engraftment will be calculated from the time of transplant and estimated by the Kaplan-Meier method.
Time to neutrophil engraftment | From the time of transplant up to 3 years
  The time to neutrophil engraftment will be calculated from the time of transplant and estimated by the Kaplan-Meier method.
Incidence of acute and chronic graft-vs.-host disease (GvHD) | Up to 3 years post-transplant
  The cumulative incidence of acute and chronic GvHD with the competing risks of relapse and death will be estimated using the method of Gooley, and the method of Fine and Gray will be used to model the association between both parameters and clinical and treatment characteristics of interest.
Incidence of relapse and non-relapse mortality | Up to 3 years post-transplant
  The cumulative incidence of non-relapse mortality and relapse will also be assessed in a competing risks framework, with similar analyses performed.
Incidence of adverse events | Up to 3 years post-transplant
  Descriptive statistics will be used to summarize adverse events. The number and proportion of subjects with treatment emergent adverse events will be reported. All other safety parameters will be summarized using descriptive statistics or frequency counts. Graphical summaries will be used where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Uday R Popat, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org